CLINICAL TRIAL: NCT04429477
Title: Assessment of Cerebral Compliance and Hemodynamics in Severe COVID-19
Brief Title: Cerebral Compliance Impairment in COVID-19
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Sergio Brasil, MD, Principal investigator, University of Sao Paulo
Other Study IDs: 31750820.1.0000.0068
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Intracranial Hypertension; Cerebral Circulatory Failure
MeSH Terms: conditions — Intracranial Hypertension | interventions — Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Cerebral compliance and hemodynamics monitoring — Noninvasive devices are been used to assess cerebral circulation and compliance.

SUMMARY:
Several recent studies point to the possibility of the new coronavirus (SARS-Cov2), which currently causes pandemic COVID-19, to infiltrate the central nervous system (CNS) and cause primary damage to neural tissues, increasing the morbidity and mortality of these patients. A pathophysiological hypothesis for insulting the CNS would be the impairment of cerebral compliance (CC), because elevation of intracranial pressure (ICP), but due to the invasive nature of the methods available for ICP evaluation, this hypothesis has so far not been verified. Recently, a noninvasive technique was developed to evaluate CC (B4C sensor), making it possible to analyse CC in patients outside the neurosurgical environment. Therefore, the main objective of this study was to assess the presence of CC impairment in patients with COVID-19, and observe potential influences of this syndrome on cerebral hemodynamics.

DETAILED DESCRIPTION:
The gravity of the disease caused by the new coronavirus 2019 (COVID-19) is predominantly harbored in severe acute respiratory syndrome (SARS), often requiring ventilatory support. However, in some cases it has been observed that the involvement of this entity is not restrict to the respiratory tract, but also to the central nervous system (CNS), heart, kidneys, intestines and testicles, or even the cross-response of the immune system with potential for Guillain-Barre and Miller-Fisher syndromes. It is not yet clear whether acute respiratory failure in patients with COVID-19 is due exclusively to pulmonary invasion or because of concurrent CNS disorders, however, as many of these patients have neurological symptoms such as headache, anosmia, paresthesia, nausea, vomiting and consciousness level alterations during the early stages of the disease, the hypothesis of this entity in promoting cerebral compliance (CC) impairment directly (i.e. encephalitis, edema or focal ischemia) or indirectly (i.e. hypoxic distress and linkage to angiotensin-converting enzyme) becomes suitable.

Intracranial pressure (ICP) monitoring is relevant in several CNS diseases with risk for critical intracranial hypertension (ICH)(10). Still, this parameter is considered in specific situations, limiting its use in neurocritical settings, especially because of the invasive nature of the monitoring techniques available. ICH has potential to compromise CC and, consequently, promote brain tissue damage. Regarding COVID-19, unless a mass effect structural damage documented by encephalic imaging is evident, there is no justification to perform a trepanation to implant an ICP monitor, hence, noninvasive techniques such as transcranial Doppler by means of cerebral hemodynamics evaluation and the novel cranial pulse detector (B4C), by means of the quantitative evaluation of the ICP curves, may play a role in this scenario.

The purpose of the present study was to evaluate CC in a set of COVID-19 patients, since implementation until withdrawal of respiratory support in ICU, to evaluate the potential persistence of CC impairment in this population. Prolonged CC impairment observation may aid decision making and targeted therapy in this population. Study design A single center, observational and prospective research was conducted including consecutive subjects in intensive care units (ICU) of the Hospital das Clínicas, São Paulo University, Brazil, with approval of local ethics committee. Our inclusion criteria regarded patients with SARS for COVID-19, under ventilatory support of any age and gender. Exclusion criteria comprehended the absence of legally authorized responsible (LAR) consent, patients without temporal acoustic window for TCD assessment, patients unable to undergo monitoring with the NICC sensor due to lesions and/or skin infections in the sensor application region, patients with head circumference smaller than 47 cm. The study protocol followed the Standards for Reporting of Diagnostic Accuracy Studies (STARD) statement.

Eligible subjects are selected by the ICU team (SF, BT, EB and LMSM) during the first three days of orotracheal intubation for CC monitoring with B4C and TCD hemodynamics evaluation once, marking the beginning of SARS. The same evaluations are repeated once again during the first three days after extubating, as a sign of recovery stage. Clinical parameters were controlled to avoid assessment bias, as systemic arterial pressure, hydric balance, presence of CNS depressors with influence on cerebrovascular hemodynamics, laboratorial partial O2 and CO2 pressures and hemoglobin, and temperature. One operator is performing TCD and B4C evaluations. Overall sample clinical condition was quantified using the simplified acute physiologic score (SAPS 3).

CC monitoring techniques Cerebral compliance was evaluated noninvasively by the cranial deformation method developed by brain4care (B4C). The B4C sensor consists of a support for a sensor bar for the detection of local cranial bone deformations adapted with deformation sensors. The detection of these deformations is obtained by a cantilever bar modeled by finite element calculations. For this bar, voltage meters are attached for deformation detection. Noninvasive contact with the skull is obtained by adequate pressure directly into the scalp by means of a pin. Variations in ICP cause deformations in the cranial bone detected by the sensor bar. The device filters, amplifies, and scans the sensor signal and sends the data to a mobile device. The method is completely non-invasive and painless. In addition, it does not interfere with any routine monitoring.

Transcranial Doppler (TCD), because it is a technique for the study of CC influences on cerebrovascular hemodynamics and vice-versa, was used to associate the information obtained by the B4C sensor. The arteries of the right and left cerebral hemispheres and the brainstem were evaluated, with Doppler colored technique with low frequency probe (2MHz) every 1 mm of arterial extension, through the temporal, orbital, suboccipital, retromastoid and submandibular windows. Arteries analyzed: proximal segments of middle, anterior and posterior cerebral arteries, paraselar and supraclinoid carotid siphons, ophthalmic, vertebral and basilar. Hemodynamic parameters of interest were mean flow velocities, peak systolic velocities, final diastolic velocities and pulsatility indexes.

Data analysis methodology Data will be analyzed obtaining a correlation coefficient and predictive ability (ROC curve) acceptable between measurements performed with the noninvasive B4C technique compared to the clinical evaluation of the patient, TCD and other available physiological parameters. To meet the objectives and goals of the study, appropriate statistical techniques will be applied. All variables will be tested for normal distribution and appropriate statistical analysis. The normality of the distribution was verified by using the Kolmogorov-Smirnov or Shapiro-Wilk test. For the demographic and basic clinical variables, descriptive data analysis was used.

The automated Brain4care Analytics system will verify all collected data by the sensor. ICP pulse wave morphology parameters such as P2/P1 ratio (P2/P1 ratio and P1 and P2 classification: P1> P2 or P2> P1) and time to peak (TTP) were obtained and stored for analysis. The calculations are performed using the mean pulse of the ICP, calculated by identifying and extracting all ICP pulses, excluding possible artifacts. The mean pulse was used to calculate the amplitudes of the P1 and P2 peaks, which were obtained by detecting the highest point of these peaks and subtracting the base value of the ICP pulse. The P2/P1 ratio was calculated by dividing the amplitude of these two points. TTP was calculated by means of standardization of the mean pulse and temporal measurement from the beginning of the pulse to its highest point (greatest amplitude).

By TCD, the first signal and elevation of ICP and CC impairment is the elevation of the pulsatility index, calculated by the following formula: PI=Sv-Dv/Mv (Sv: systolic velocity, Dv: diastolic velocity and Mv: mean flow velocity), since excluded confounding factors such as distal stenosis of the cranial arteries, use of barbiturate in infusion pump, dehydration, sepsis, aortic or microvascular cerebral valve failure (microangiopathy) for example. Later, in situations of more severe intracranial hypertension, tissue tension is translated by TCD as sharper systolic peaks, observed by the suppression of the second systolic peak (sys2).

ELIGIBILITY:
Inclusion Criteria:

* patients with SARS for COVID-19, under ventilatory support of any age and gender

Exclusion Criteria:

* the absence of legally authorized responsible (LAR) consent,
* patients without temporal acoustic window for TCD assessment,
* patients unable to undergo monitoring with the NICC sensor due to lesions and/or skin infections in the sensor application region,
* patients with head circumference smaller than 47 cm.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects were selected by the ICU team during the first three days of orotracheal intubation for CC monitoring with B4C and TCD hemodynamics evaluation once, marking the beginning of SARS. The same evaluations were repeated once again during the first three days after orotracheal tube withdrawal, as a sign of recovery stage. Clinical parameters were controlled to avoid assessment bias, as systemic arterial pressure, hydric balance, presence of CNS depressors with influence on cerebrovascular hemodynamics, laboratorial partial O2 and CO2 pressures and hemoglobin, and temperature. One operator is performing TCD and B4C evaluations. Overall sample clinical condition is quantified using the simplified acute physiologic score (SAPS 3). Each subject undergone a skull CT scan in order to exclude a mass effect lesion not related to COVID-19.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Detection of cerebral compliance impairment by the B4C sensor | During critical care, around 15 days/patient
  Observe alteration in cerebral compliance due to potential intracranial hypertension during severe COVID-19. This situation is indicated when the relation P2/P1 given by the B4C sensor is >1.
Detection of cerebral hemodynamics impairment by transcranial Doppler | During critical care, around 15 days/patient
  Observe disturbances in cerebral circulation during severe COVID-19, given by blood flow velocities in middle cerebral arteries (with normal range 40-70 cm/s) and the pulsatility index (normal <1.2) calculated by transcranial Doppler.

SECONDARY OUTCOMES:
Calculate mortality in this population | 3 months
  Observe whether disturbances in cerebral compliance and hemodynamics assessed in this population is significantly associated with higher mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li YC, Bai WZ, Hashikawa T. The neuroinvasive potential of SARS-CoV2 may play a role in the respiratory failure of COVID-19 patients. J Med Virol. 2020 Jun;92(6):552-555. doi: 10.1002/jmv.25728. Epub 2020 Mar 11. PMID 32104915
- [Background] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Background] Needham EJ, Chou SH, Coles AJ, Menon DK. Neurological Implications of COVID-19 Infections. Neurocrit Care. 2020 Jun;32(3):667-671. doi: 10.1007/s12028-020-00978-4. PMID 32346843
- [Background] Bridwell R, Long B, Gottlieb M. Neurologic complications of COVID-19. Am J Emerg Med. 2020 Jul;38(7):1549.e3-1549.e7. doi: 10.1016/j.ajem.2020.05.024. Epub 2020 May 16. PMID 32425321
- [Background] Niazkar HR, Zibaee B, Nasimi A, Bahri N. The neurological manifestations of COVID-19: a review article. Neurol Sci. 2020 Jul;41(7):1667-1671. doi: 10.1007/s10072-020-04486-3. Epub 2020 Jun 1. PMID 32483687
- [Background] Wu Y, Xu X, Chen Z, Duan J, Hashimoto K, Yang L, Liu C, Yang C. Nervous system involvement after infection with COVID-19 and other coronaviruses. Brain Behav Immun. 2020 Jul;87:18-22. doi: 10.1016/j.bbi.2020.03.031. Epub 2020 Mar 30. PMID 32240762
- [Background] Delanghe JR, Speeckaert MM, De Buyzere ML. The host's angiotensin-converting enzyme polymorphism may explain epidemiological findings in COVID-19 infections. Clin Chim Acta. 2020 Jun;505:192-193. doi: 10.1016/j.cca.2020.03.031. Epub 2020 Mar 24. No abstract available. PMID 32220422
- [Background] Kochanek PM, Tasker RC, Carney N, Totten AM, Adelson PD, Selden NR, Davis-O'Reilly C, Hart EL, Bell MJ, Bratton SL, Grant GA, Kissoon N, Reuter-Rice KE, Vavilala MS, Wainwright MS. Guidelines for the Management of Pediatric Severe Traumatic Brain Injury, Third Edition: Update of the Brain Trauma Foundation Guidelines, Executive Summary. Neurosurgery. 2019 Jun 1;84(6):1169-1178. doi: 10.1093/neuros/nyz051. PMID 30822776
- [Background] Frigieri G, Andrade RAP, Dias C, Spavieri DL Jr, Brunelli R, Cardim DA, Wang CC, Verzola RMM, Mascarenhas S. Analysis of a Non-invasive Intracranial Pressure Monitoring Method in Patients with Traumatic Brain Injury. Acta Neurochir Suppl. 2018;126:107-110. doi: 10.1007/978-3-319-65798-1_23. PMID 29492543
- [Background] Vilela GH, Cabella B, Mascarenhas S, Czosnyka M, Smielewski P, Dias C, Cardim DA, Mascarenhas YM, Wang CC, Andrade R, Tanaka K, Lopes LS, Colli BO. Validation of a New Minimally Invasive Intracranial Pressure Monitoring Method by Direct Comparison with an Invasive Technique. Acta Neurochir Suppl. 2016;122:97-100. doi: 10.1007/978-3-319-22533-3_19. PMID 27165885
- [Background] Cabella B, Vilela GH, Mascarenhas S, Czosnyka M, Smielewski P, Dias C, Cardim DA, Wang CC, Mascarenhas P, Andrade R, Tanaka K, Silva Lopes L, Colli BO. Validation of a New Noninvasive Intracranial Pressure Monitoring Method by Direct Comparison with an Invasive Technique. Acta Neurochir Suppl. 2016;122:93-6. doi: 10.1007/978-3-319-22533-3_18. PMID 27165884
- [Background] Schaafsma A. A new method for correcting middle cerebral artery flow velocity for age by calculating Z-scores. J Neurosci Methods. 2018 Sep 1;307:1-7. doi: 10.1016/j.jneumeth.2018.06.009. Epub 2018 Jun 18. PMID 29920296
- [Background] Schaafsma A. Improved parameterization of the transcranial Doppler signal. Ultrasound Med Biol. 2012 Aug;38(8):1451-9. doi: 10.1016/j.ultrasmedbio.2012.03.016. Epub 2012 May 12. PMID 22579541